CLINICAL TRIAL: NCT06533098
Title: Multicenter, Open-Label, Randomized Study of Nipocalimab or Intravenous Immunoglobulin (IVIG) in Pregnancies At Risk of Fetal and Neonatal Alloimmune Thrombocytopenia (FNAIT)
Brief Title: A Study of Nipocalimab or Intravenous Immunoglobulin (IVIG) in Pregnancies At Risk of Fetal and Neonatal Alloimmune Thrombocytopenia (FNAIT)
Acronym: FREESIA-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80202135FNAIT3003; 80202135FNAIT3003 (Other: Janssen Research & Development, LLC); 2023-509434-19-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thrombocytopenia, Neonatal Alloimmune
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune | interventions — Immunoglobulins, Intravenous; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Nipocalimab (Experimental): Maternal participants with alloantibodies against HPA-1a and/or HPA-5b will be randomized to receive nipocalimab starting at gestational age (GA) week 13 to 18 until before delivery.
  Interventions: Drug: Nipocalimab
- Arm 2: Intravenous Immunoglobins (IVIG) (Experimental): Maternal participants with alloantibodies against HPA-1a and/or HPA-5b will be randomized to receive IVIG from GA week 12 for high-risk pregnancies or GA week 20 for standard-risk pregnancies. Additionally, prednisone will be added per study protocol. Participants will be gradually tapered off prednisone after delivery as per investigator judgement or maternal participant tolerance.
  Interventions: Drug: Intravenous immunoglobulins (IVIG); Drug: Prednisone

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered intravenously.
  Other Names: JNJ-80202135; JNJ-86507083
  Arms: Arm 1: Nipocalimab
Drug: Intravenous immunoglobulins (IVIG) — IVIG will be administered intravenously.
  Arms: Arm 2: Intravenous Immunoglobins (IVIG)
Drug: Prednisone — Prednisone will be administered orally.
  Arms: Arm 2: Intravenous Immunoglobins (IVIG)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of nipocalimab in reducing the risk of severe fetal and neonatal alloimmune thrombocytopenia (FNAIT).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and an estimated gestational age from week 13 to 18 at visit 1
* Has a history of greater than or equal to (>=) 1 prior pregnancy with FNAIT based on medical records including: a) neonatal platelet count less than (<) 150*10^9/Liter with no fetal/neonatal intracranial hemorrhage (ICH) or severe fetal/neonatal hemorrhage (standard-risk) OR b) fetus/neonate with ICH or severe hemorrhage in a fetus/neonate (high-risk)
* Current pregnancy with presence of maternal anti-HPA-1a and/or anti-HPA-5b alloantibody and positive fetal HPA-1a and/or HPA-5b genotype as confirmed by cell-free fetal DNA in maternal blood
* Health status considered stable by the investigator based on physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening
* For maternal participant and neonate/infant, willing to forego participation in another clinical study of an investigational therapy until the last follow-up visit

Exclusion Criteria:

* Currently pregnant with multiple gestations (twins or more)
* History of severe preeclampsia in a previous pregnancy
* History of myocardial infarction, unstable ischemic heart disease, or stroke
* Known allergies, hypersensitivity, or intolerance to nipocalimab or its excipients, to IVIG or to prednisone
* Has any confirmed or suspected clinical immunodeficiency syndrome or has a family history of congenital or hereditary immunodeficiency unless confirmed absent in the participant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-12-05 (Estimated)

PRIMARY OUTCOMES:
Fetus/Neonate with Outcome of Death or Adjudicated Severe Bleeding or Platelet Count Less Than (<) 30*10^9/L | Up to 1 Week post birth
  Outcome of fetus/neonate death or adjudicated severe bleeding up to the first week post birth or platelet count <30*10^9/L will be reported.

SECONDARY OUTCOMES:
Platelet Count at Birth in a Neonate | At birth
  Platelet count at birth in a neonate will be reported.
Neonate/Fetus with Outcome of Death | Up to 1 Week post birth
  Fetus/neonate with outcome of death will be reported.
Neonate with Platelet Count at Birth <10*10^9/L | At birth
  Platelet count at birth <10*10^9/L in a neonate will be reported.
Neonate with Platelet Count at Birth <30*10^9/L | At birth
  Platelet count at birth <30*10^9/L in a neonate will be reported.
Neonate with Platelet Count at Birth <50*10^9/L | At birth
  Platelet count at birth <50*10^9/L in a neonate will be reported.
Neonate with Platelet Count at Birth <150*10^9/L | At birth
  Platelet count at birth <150*10^9/L in a neonate will be reported.
Nadir Platelet Count in a Neonate | Up to 1 Week post birth
  Nadir platelet count in a neonate will be reported.
Neonate Requiring Platelet Transfusion | Up to 1 Week post birth
  Neonate who require at least one platelet transfusion will be reported.
Number of Platelet Transfusions in Neonate | Up to 1 Week post birth
  Number of platelet transfusions per neonate will be reported.
Number of Donor Exposures for Platelet Transfusions in Neonate | Up to 1 Week post birth
  Number of donor exposures for a neonate who received at least one platelet transfusion will be reported.
Neonate/Fetus With Adjudicated Bleeding | Up to 1 Week post birth
  Neonate/Fetus with adjudicated bleeding will be reported.
Neonate Requiring Postnatal Intravenous Immunoglobulin (IVIG) for the Treatment of Thrombocytopenia | Up to 1 Week post birth
  Neonate requiring IVIG for the treatment of thrombocytopenia will be reported.
Maternal Participant with Treatment-Emergent Adverse Events (TEAE), Serious Adverse Events (SAE) and Adverse Event of Special Interest (AESI) | Up to Week 24
  Maternal participant with TEAE, SAE and AESI will be reported. An Adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study.
Maternal Participant with TEAE Leading to Discontinuation of Study Intervention | Up to Week 24
  Maternal participant with TEAE leading to discontinuation of study intervention will be reported.
Neonate/Infant With TEAE, SAE and AESI | From Day of birth to Week 104
  Neonate/infant with TEAE, SAE and AESI will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study.
Fetus/Neonate with a TEAE of Bleeding | From Day of birth to Week 104
  Fetus/Neonate with a TEAE of bleeding will be reported.
Neonate with a TEAE of Infection | From Day of birth to Week 104
  Neonate with a TEAE of infection will be reported.
Bayley Scales Assessment for Infant Development | At Week 52 and Week 104
  The Bayley Scales of infant development is considered the standard assessment of early child development and includes cognition, language, motor skills, social emotional, and adaptive behavior will be reported. The Bayley Scales are reference standards that measure infant and toddler development in five areas: cognition, language, motor skills, social-emotional and adaptive behavior. The cognition, language and motor skills scales are directly administered to the infant, while social-emotional, and adaptive behavior scales are caregiver questionnaires. The scores are standardized using norm reference samples with representative demographics and age adjusted for prematurity. Higher scores in the Bayley Scales indicate better outcomes.
Maternal Participants with Incidence of Antibodies to Nipocalimab | Up to Week 4
  Incidence of antibodies to nipocalimab including neutralizing antibodies in maternal serum during pregnancy and postpartum will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (20):
- United States (6):
  - UC Davis School of Medicine, Sacramento, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Advocate Children's Hospital, Park Ridge, Illinois
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Medical University Vienna, Vienna
- Germany (4):
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Jena, Jena
  - Universitaetsklinikum Tuebingen, Tübingen
- Leiden University Medical Center, Leiden, Netherlands
- Poland (3):
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Instytut Matki i Dziecka, Warsaw
  - Panstwowy Instytut Medyczny MSWiA w Warszawie, Warsaw
- United Kingdom (4):
  - Birmingham Women's Hospital, Birmingham
  - Liverpool Women's NHS Foundation Trust - Liverpool Women's Hospital, Liverpool
  - Queen Charlotte's and Chelsea Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Bussel J, Stegmann B, Baker P, Oey A, Jiang Y, Zaha R, Van Valkenburgh H, Keshinro B. Design of a Phase 3, Multicenter, Randomized, Open-Label Study of Nipocalimab or IVIG and Prednisone in Pregnancies at Risk for Fetal and Neonatal Alloimmune Thrombocytopenia. Am J Perinatol. 2025 Dec 12. doi: 10.1055/a-2753-9323. Online ahead of print. PMID 41290206